CLINICAL TRIAL: NCT06886230
Title: Assessing The Safety and Efficacy of Ondansetron, Dexamethasone, and Their Combined Regimen in Managing Post Operative Nausea and Vomiting: A Randomized Controlled Trial
Brief Title: Ondansetron vs. Dexamethasone for Postoperative Nausea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hafiz Muhammad Hamza (Other)
Collaborators: Federal Government Polyclinic (Postgraduate Medical Institute) (Other)
Responsible Party: Sponsor-Investigator, Hafiz Muhammad Hamza, House Officer, Foundation University School of Health Sciences, Federal Government Polyclinic (Postgraduate Medical Institute)
Organization: Federal Government Polyclinic (Postgraduate Medical Institute) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FGPC.1/12/2024 E-Committee
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
Keywords: nausea; vomiting; PONV; randomized controlled trial; ondansetron; dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Saline Solution; Sodium Chloride; Ondansetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: This study follows a randomized, parallel-group, single blinded placebo-controlled interventional design to assess the efficacy and safety of Ondansetron, Dexamethasone, and their combination in preventing postoperative nausea and vomiting (PONV).
Who Masked: Participant
Masking Description: This study will be single-blinded, meaning that the patients will not be aware of their assigned treatment group, but the healthcare provider administering the medication will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Placebo Group (Control) (Placebo Comparator): Patients in this group will receive a placebo (normal saline) intravenously before surgery. This group serves as a control to compare the efficacy and safety of the active treatment regimens.
  Interventions: Drug: Placebo (Normal Saline)
- Arm 2: Ondansetron Group (Active Comparator): Patients in this group will receive a single dose of Ondansetron 4 mg IV before surgery. Ondansetron is a 5-hydroxytryptamine type 3 receptors antagonist commonly used for postoperative nausea and vomiting prevention.
  Interventions: Drug: Ondansetron (Zofran)
- Arm 3: Dexamethasone Group (Active Comparator): Patients in this group will receive a single dose of Dexamethasone 8 mg IV before surgery. Dexamethasone is a corticosteroid that has been shown to reduce postoperative nausea and vomiting.
  Interventions: Drug: Dexamethasone
- Arm: 4 Combination Therapy Group (Active Comparator): Patients in this group will receive a combination of Ondansetron 4 mg IV and Dexamethasone 8 mg IV before surgery. The combination therapy is expected to have an additive effect in reducing PONV.
  Interventions: Drug: Ondansetron (Zofran); Drug: Dexamethasone

INTERVENTIONS:
Drug: Placebo (Normal Saline) — Patients in this group will receive an intravenous (IV) injection of normal saline before surgery. This serves as a control group to compare the efficacy of active treatment groups in preventing postoperative nausea and vomiting.
  Other Names: Saline Injection; Inert Solution
  Arms: Arm 1: Placebo Group (Control)
Drug: Ondansetron (Zofran) — Patients in this group will receive a single intravenous (IV) dose of Ondansetron 4 mg before surgery. Ondansetron is a selective 5-HT3 receptor antagonist commonly used to prevent nausea and vomiting associated with anesthesia and surgery.
  Other Names: Zofran; Ondem; Emeset
  Arms: Arm 2: Ondansetron Group; Arm: 4 Combination Therapy Group
Drug: Dexamethasone — Patients in this group will receive a single intravenous (IV) dose of Dexamethasone 8 mg before surgery. Dexamethasone is a corticosteroid with anti-inflammatory properties that has been shown to reduce the incidence of PONV by modulating inflammatory pathways and neuroreceptor activity.
  Other Names: Decadron; Dexasone
  Arms: Arm 3: Dexamethasone Group; Arm: 4 Combination Therapy Group

SUMMARY:
This randomized controlled trial aims to evaluate the safety and efficacy of Ondansetron, Dexamethasone, and their combination in managing postoperative nausea and vomiting (PONV) in patients undergoing surgery under anesthesia. A total of 100 patients will be randomized into four groups: Placebo, Ondansetron, Dexamethasone, and Ondansetron-Dexamethasone combination. The primary outcome will be the incidence of PONV within 24 hours post-surgery, while secondary outcomes include severity of symptoms, need for rescue medication, adverse effects, and patient satisfaction.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common and distressing complication following surgery, affecting patient recovery and satisfaction. This study aims to compare the safety and effectiveness of Ondansetron, Dexamethasone, and their combination for PONV prevention.

The study will be conducted as a randomized, controlled trial at Federal Polyclinic Hospital Islamabad over four months. A total of 100 adult patients undergoing elective surgery under anesthesia will be enrolled and randomly allocated into one of four groups (n=25 each):

Placebo group - Receives no prophylactic antiemetic treatment. Ondansetron group - Receives 4 mg IV Ondansetron before surgery. Dexamethasone group - Receives 8 mg IV Dexamethasone before surgery. Ondansetron-Dexamethasone group - Receives 4 mg IV Ondansetron + 8 mg IV Dexamethasone before surgery.

Methodology:

Patients will be assessed at multiple time points (2, 4, 6, 12, and 24 hours postoperatively) for PONV incidence and severity, along with the need for rescue medication. Side effects such as headache, dizziness, hypertension, and hyperglycemia will also be monitored.

Statistical Analysis:

Data will be analyzed using chi-square tests and ANOVA to compare outcomes across treatment groups. A p-value < 0.05 will be considered statistically significant.

This study will help determine the most effective and safest antiemetic regimen, guiding clinical decision-making for better PONV management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) scheduled for elective surgery under anesthesia.
* Patients at moderate to high risk for postoperative nausea and vomiting (PONV), as determined by an Apfel risk score ≥2.
* Patients able to provide informed consent or have a legally authorized representative provide consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to Ondansetron, Dexamethasone, or any of their components.
* History of significant adverse reactions to previous PONV prophylaxis with Ondansetron or Dexamethasone.
* Pre-existing conditions or medications contraindicating the use of Ondansetron or Dexamethasone, e.g. QT prolongation or severe cardiac arrhythmias (e.g., torsades de pointes, congenital long QT syndrome), Uncontrolled hypertension (for Dexamethasone use), Severe hepatic impairment (Child-Pugh C) or end-stage renal disease, Uncontrolled diabetes mellitus (due to Dexamethasone-induced hyperglycemia).
* Patients with active malignancy undergoing chemotherapy or radiotherapy.
* Pregnant or lactating women (unless safety in this population is specifically being studied).
* Chronic opioid users (≥3 months of continuous opioid use), as this may alter PONV risk and response to prophylaxis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | 24 hours
  Defined as the presence of nausea and/or vomiting at any assessment time point (recovery, 2, 4, 6, 12, and 24 hours postoperatively).
  Comparison of postoperative nausea and vomiting incidence between the Ondansetron-Dexamethasone and Ondansetron groups.
  The need for rescue antiemetic administration as an indicator of postoperative nausea and vomiting severity.

SECONDARY OUTCOMES:
Severity of Postoperative Nausea and Vomiting (Postoperative Nausea and Vomiting Impact Scale Score) | 24 hours
  Assessment of the frequency, severity, and impact of nausea and vomiting on daily activities and quality of life.
  Measured using patient-reported responses to the Postoperative Nausea and Vomiting Impact Scale.
  Scoring Range: 0 to 6 Minimum Score (0): No impact of nausea or vomiting Maximum Score (6): Severe impact on daily activities Interpretation: Higher scores indicate a worse outcome, with greater severity and impact of PONV.
Postoperative Pain Scores (Visual Analog Scale Score) | 24 hours
  Pain intensity recorded at recovery, 2, 6 and 24 hours postoperatively using the Visual Analog Scale. A 10-point scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate greater pain severity.
  Comparison of pain levels between the two groups to determine any analgesic effects of dexamethasone.
Need for Rescue Medication | 24 hours
  Frequency and timing of rescue antiemetic administration in both groups. Determines the effectiveness of the interventions in controlling postoperative nausea and vomiting.
Adverse Effects of Medications | 24 hours
  Frequency of ondansetron-related side effects: headache, dizziness, constipation, diarrhea, fatigue, allergic reactions.
  Frequency of dexamethasone-related side effects: increased appetite, insomnia, mood changes, fluid retention, hypertension, hyperglycemia.
Satisfaction with Postoperative Nausea and Vomiting Management | 24 hours
  Patient-reported satisfaction levels with nausea and vomiting management, measured using the satisfaction scale in the questionnaire.
  Each response is scored on a 5-point Likert scale, where:
  1. = Very dissatisfied (minimum score)
  2. = Somewhat dissatisfied
  3. = Neutral
  4. = Somewhat satisfied
  5. = Very satisfied (maximum score) The total score ranges from 5 (minimum satisfaction) to 25 (maximum satisfaction), with higher scores indicating better patient satisfaction.
Apfel Score: Risk Assessment for Postoperative Nausea and Vomiting (PONV) | 24 hours
  Apfel Score Components (Each Risk Factor = 1 Point) Female gender → (Yes = 1 point, No = 0 points) History of postoperative nausea and vomiting or motion sickness → (Yes = 1 point, No = 0 points) Non-smoker → (Yes = 1 point, No = 0 points) Planned use of postoperative opioid analgesia → (Yes = 1 point, No = 0 points) Higher Apfel Scores indicate an increased risk of postoperative nausea and vomiting.
Heart Rate | 24 hours
  Heart rate (beats per minute) will be continuously monitored and recorded at predefined intraoperative and postoperative time points to assess hemodynamic stability and detect potential bradycardia or tachycardia.
Blood Pressure | 24 hours
  Systolic and diastolic blood pressure (measured in mmHg) will be recorded at regular intraoperative and postoperative intervals to monitor hemodynamic stability and detect episodes of hypotension or hypertension.
Respiratory Rate | 24 hours
  Respiratory rate (measured in breaths per minute) will be monitored intraoperatively and postoperatively to evaluate respiratory function and detect potential respiratory depression or distress.
Oxygen Saturation | 24 hours
  Oxygen saturation levels (SpO₂, measured as a percentage) will be continuously monitored throughout the intraoperative and postoperative periods to assess respiratory function and detect hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Ullah Khan, Consultant surgery, HOD, Principal Investigator — Federal Government Polyclinic (Postgraduate Medical Institute)
Locations (1):
- Federal Government Polyclinic (Postgraduate Medical Institute), Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no final decision has been made regarding the sharing of individual participant data (IPD). Data sharing will be considered based on future research needs, ethical guidelines, and institutional policies. Any decision to share IPD will be made in compliance with data protection regulations and patient confidentiality standards.

REFERENCES:
- [Background] Bhattarai B, Shrestha S, Singh J. Comparison of ondansetron and combination of ondansetron and dexamethasone as a prophylaxis for postoperative nausea and vomiting in adults undergoing elective laparoscopic surgery. J Emerg Trauma Shock. 2011 Apr;4(2):168-72. doi: 10.4103/0974-2700.82200. PMID 21769200
- [Background] Thanuja IL, Parida S, Mishra SK, Badhe AS. Effect of combinations of dexamethasone-ondansetron and dexamethasone-ondansetron-aprepitant versus aprepitant alone for early postoperative nausea and vomiting after day care gynaecological laparoscopy: A randomised clinical trial. Indian J Anaesth. 2021 Jun;65(6):465-470. doi: 10.4103/ija.IJA_119_21. Epub 2021 Jun 22. PMID 34248190
- [Background] Bilgen S, Kizilcik N, Haliloglu M, Yildirim G, Kaspar EC, Koner O. Effect of the Dexamethasone-Ondansetron Combination Versus Dexamethasone-Aprepitant Combination to Prevent Postoperative Nausea and Vomiting. Turk J Anaesthesiol Reanim. 2018 Sep;46(5):373-380. doi: 10.10.5152/TJAR.2018.53179. Epub 2018 Sep 4. PMID 30263861
- See also: Dexamethasone, ondansetron, and their combination and postoperative nausea and vomiting in children undergoing strabismus surgery: a meta-analysis of randomized controlled trials — https://pubmed.ncbi.nlm.nih.gov/24612183/